CLINICAL TRIAL: NCT04338685
Title: A First In Human, Open Label, Dose Escalation Phase I Study Evaluating Safety, Pharmacokinetics, Pharmacodynamics, And Preliminary Clinical Activity Profile Of Single Agent RO7119929 (TLR7 Agonist) Administered Orally To Participants With Unresectable Advanced Or Metastatic Hepatocellular Carcinoma, Biliary Tract Cancer, Or Solid Tumors With Hepatic Metastases
Brief Title: A Study Evaluating Safety, Pharmacokinetics, Pharmacodynamics, And Clinical Activity Of RO7119929 (TLR7 Agonist) In Participants With Unresectable Advanced Or Metastatic Hepatocellular Carcinoma, Biliary Tract Cancer, Or Solid Tumors With Hepatic Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WP41377
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Carcinoma, Hepatocellular; Biliary Tract Cancer; Secondary Liver Cancer; Liver Metastases
Keywords: TLR7 Agonist
MeSH Terms: conditions — Carcinoma, Hepatocellular; Biliary Tract Neoplasms | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Open label, multi-center, single-arm, multiple-ascending dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part A1-1 mg RO7119929 (Experimental): Participants received 1mg RO7119929 every week in 3-week cycles.
  Interventions: Drug: RO7119929
- Part A1-3 mg RO7119929 (Experimental): Participants received 4 mg RO7119929 every week in 3-week cycles
  Interventions: Drug: RO7119929
- Part A1 - 6 mg RO7119929 (Experimental): Participants received 6 mg RO7119929 every week in 3-week cycles
  Interventions: Drug: RO7119929
- Part A1 -9 mg RO7119929 (Experimental): Participants received 9 mg RO7119929 every week in 3-week cycles
  Interventions: Drug: RO7119929
- Part B1-5 mg RO7119929 (Experimental): Participants with both available and evaluable tumor biopsy samples received 5 mg RO7119929 on Cycle 1 Day 1 to month 12
  Interventions: Drug: RO7119929
- Part A2- 2/5/5 mg RO7119929 (Experimental): Participants received RO7119929 QW with step-up dosing of 2/5/5 mg during Cycle 1.
  Interventions: Drug: RO7119929
- Part A2- 2/5/6 mg RO7119929 (Experimental): Participants received RO7119929 QW with step-up dosing of 2/5/6 mg during Cycle 1.
  Interventions: Drug: RO7119929
- Part A3-4 mg RO7119929 (Experimental): Participants received tocilizumab pre-treatment on Cycle 1 Day 1, approximately 2 hours prior to RO7119929 administration and 4 mg RO7119929 every week in 3-week cycles
  Interventions: Drug: RO7119929; Drug: Tocilizumab

INTERVENTIONS:
Drug: RO7119929 — RO7119929 will be administered orally as a capsule
Drug: Tocilizumab — Tocilizumab will be administered in case of severe steroid-refractory cytokine release syndrome.
  Tocilizumab will be administered as concentrate for solution for IV infusion at a dose: for participants > 30 kg: 8 mg/kg, for participants < 30 kg: 12mg/kg IV
  Other Names: Actemra
  Arms: Part A3-4 mg RO7119929

SUMMARY:
Phase I study of RO7119929 given orally to participants with unresectable advanced or metastatic primary liver cancers and other solid tumors with predominant liver involvement. The primary objective of the study is to explore the safety and to determine the maximum tolerated dose (MTD) and/or optimal biologic dose (OBD) of RO7119929 as single agent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of one of the following: unresectable advanced or metastatic HCC (including fibrolamellar HCC) not amenable to a curative treatment approach, unresectable advanced or metastatic intrahepatic or perihilar (Klatskin) BTC not amenable to a curative treatment approach, extrahepatic BTC or gallbladder cancer infiltrating the liver or metastasized into the liver with predominant liver disease, not amenable to a curative treatment approach, metastasized colorectal cancer (CRC), pancreatic ductal adenocarcinoma (PDAC), Gastric cancer (GC), renal cell carcinoma (RCC), triple negative breast cancer (TNBC), cutaneous melanoma, or ocular melanoma with predominant liver disease not amenable to a curative treatment approach. Participants with other solid tumors with predominant liver disease not amenable to a curative treatment approach might be enrolled after Sponsor approval
* Measurable disease with at least one measurable locally untreated liver lesion, as defined by RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate hematologic and major organ functions
* Participants for which there is no available standard therapy likely to confer clinical benefit, or participants who are not candidates for such available therapy
* Life expectancy of ≥12 weeks, approximated with Royal Marsden Hospital score 0-1 or Gustave Roussy Immune (GRIm) score 0-1. Participants with a Royal Marsden Hospital or GRIm score of ≥2 and a life expectancy of ≥12 weeks according to the investigator's clinical judgement may be enrolled after Medical Monitor approval has been obtained.
* For participants with HCC: Child-Pugh score of A6 or better

Exclusion Criteria:

* History or clinical evidence of central nervous system (CNS) primary tumors or metastases including leptomeningeal metastases, unless they have been previously treated, are asymptomatic, and have had no requirement for steroids or enzyme-inducing anticonvulsants in the last 14 days prior to Screening
* Evidence of any extra-hepatic primary tumor or metastasis requiring prompt medical intervention
* Receipt of prior therapy with a TLR7/8/9 agonist and/or IFN-alpha
* Prior chemotherapy, antibody, or other registered or experimental cancer treatment within 3 weeks of study Cycle 1 Day 1. Specifically, no CPI antibody is allowed to be administered within 6 weeks of study Cycle 1 Day 1
* Receipt of investigational agent for any other indication within 3 weeks of dosing
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment
* Local therapy to liver (e.g. radiofrequency ablation, percutaneuous ethanol or acetic acid injection, cryoablation, high-intensity focused ultrasound, transarterial chemoembolization, and transarterial embolization) within 3 weeks prior to initiation of study treatment, radioembolization within 3 months prior to initiation of study treatment, or non-recovery from side effects of such procedure
* Treatment-related toxicities from prior cancer therapy that have not resolved to </= Grade 1 CTC AE prior to study treatment with the exception of the following Grade 2 toxicities:

alopecia, peripheral neuropathy, any laboratory changes that still lie within the inclusion criteria defined above

* History of other malignancy within 2 years; exception for ductal carcinoma in situ not requiring chemotherapy, low grade cervical intraepithelial neoplasia (CIN), nonmelanoma skin cancer, low grade localized prostate cancer (Gleason score < Grade 7), or optimally treated Stage 1 uterine cancer.
* Active or history of immunologic-mediated disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren's syndrome or Guillain-Barré syndrome
* Known active or uncontrolled bacterial, viral, fungal, mycobacterial, parasitic, or other infection.
* Ascites, pleural effusion, or pericardial effusion requiring medical intervention within 12 months prior to study entry.
* History of human immunodeficiency virus (HIV) infection
* Active hepatitis B virus (HBV) infection
* Coinfection of HBV and hepatitis C virus (HCV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- City of Hope Cancer Center, Duarte, California, United States
- Rigshospitalet; Onkologisk Klinik, København Ø, Denmark
- Queen Mary Hospital; Dept of Medicine, Hong Kong, Hong Kong
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (3):
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron; Oncology, Barcelona
  - Clinica Universidad de Navarra Madrid; Servicio de Oncología, Madrid
- Taiwan (2):
  - National Taiwan Uni Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At Cycle 1 Day 1, Cycle 1 Day 8, and Cycle 1 Day 15, the participant were pre-medicated with 500 mL of crystalloid fluid and 500-1000 mg paracetamol orally (PO) or intravenously (IV) at the time of RO7119929 administration (± 30 minutes), followed by 500-1000 mg paracetamol PO or IV 4-6 hours after first drug administration. If no cytokine release syndrome (CRS) is observed, no further premedication was foreseen beyond Cycle 1.
Groups:
- Part A1-3 mg RO7119929: Participants received 3 mg RO7119929 every week in 3-week cycles.
- Part A1 -4 mg RO7119929: Participants received 4 mg RO7119929 every week in 3-week cycles
Period: Overall Study
Arm/Group | Part A1-1 mg RO7119929 | Part A1-3 mg RO7119929 | Part A1 -4 mg RO7119929 | Part A1 - 6 mg RO7119929 | Part A1 -9 mg RO7119929 | Part B1-5 mg RO7119929 | Part A2- 2/5/5 mg RO7119929 | Part A2- 2/5/6 mg RO7119929 | Part A3-4 mg RO7119929
Started | 4 | 6 | 3 | 10 | 4 | 18 | 4 | 5 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 6 | 3 | 10 | 4 | 18 | 4 | 5 | 1
Not completed — Death | 3 | 4 | 2 | 4 | 4 | 8 | 1 | 0 | 0
Not completed — Study terminated by Sponsor | 0 | 0 | 1 | 4 | 0 | 5 | 2 | 4 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 2 | 0 | 5 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A1-1 mg RO7119929 | Part A1-3 mg RO7119929 | Part A1 -4 mg RO7119929 | Part A1 - 6 mg RO7119929 | Part A1 -9 mg RO7119929 | Part B1-5 mg RO7119929 | Part A2- 2/5/5 mg RO7119929 | Part A2- 2/5/6 mg RO7119929 | Part A3-4 mg RO7119929 | Total
Number analyzed (Participants) | 4 | 6 | 3 | 10 | 4 | 18 | 4 | 5 | 1 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 1 | 7 | 1 | 14 | 3 | 5 | 1 | 41
  >=65 years | 1 | 0 | 2 | 3 | 3 | 4 | 1 | 0 | 0 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.0 (5.0) | 57.5 (5.0) | 69.3 (10.8) | 55.9 (12.6) | 62.8 (16.0) | 57.6 (9.8) | 55.3 (10.7) | 53.0 (10.3) | 68.0 (NA) — Only 1 participant analyzed, SD cannot be calculated. | 58.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 5 | 0 | 14 | 0 | 1 | 0 | 23
  Male | 3 | 5 | 2 | 5 | 4 | 4 | 4 | 4 | 1 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 6 | 3 | 10 | 4 | 18 | 4 | 5 | 1 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 2 | 4 | 3 | 7 | 2 | 3 | 0 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 2 | 1 | 6 | 1 | 11 | 2 | 2 | 1 | 27
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: A DLT is defined as a clinically significant AE (classified according to the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v.5.0) or significant laboratory abnormality 1) occurring during an assessment period of 21 days or 28 days after first dose of study treatment, respectively, and 2) is not attributed to disease progression, concomitant illness or another clearly identifiable cause.
Time Frame: Baseline up to approximately 14 months
Measure: Number; unit: Participants
Arm/Group | Part A1-1 mg RO7119929 | Part A1-3 mg RO7119929 | Part A1 -4 mg RO7119929 | Part A1 - 6 mg RO7119929 | Part A1 -9 mg RO7119929 | Part B1-5 mg RO7119929 | Part A2- 2/5/5 mg RO7119929 | Part A2- 2/5/6 mg RO7119929 | Part A3-4 mg RO7119929
Number analyzed (Participants) | 4 | 6 | 3 | 10 | 4 | 18 | 4 | 5 | 1
Participants | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Events (AEs) According To NCI CTCAE v5.0
Description: An Adverse Event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Baseline up to approximately 14 months
Measure: Number; unit: Participants
Arm/Group | Part A1-1 mg RO7119929 | Part A1-3 mg RO7119929 | Part A1 -4 mg RO7119929 | Part A1 - 6 mg RO7119929 | Part A1 -9 mg RO7119929 | Part B1-5 mg RO7119929 | Part A2- 2/5/5 mg RO7119929 | Part A2- 2/5/6 mg RO7119929 | Part A3-4 mg RO7119929
Number analyzed (Participants) | 4 | 6 | 3 | 10 | 4 | 18 | 4 | 5 | 1
Participants
  Participants with Adverse Events | 3 | 6 | 3 | 10 | 3 | 18 | 4 | 5 | 1
  Participants with Serious Adverse Events | 1 | 2 | 2 | 4 | 4 | 11 | 1 | 2 | 0

3. Secondary Outcome: Maximum Concentration (Cmax) for RO7119929 Following Administration of RO7119929
Time Frame: Cycle 1, after 1st dose, Cycle 2, after 4th dose (Each cycle is 21 days)
Population: Participants in 9 mg cohort were excluded from the Cycle 2 analysis (2 discontinued the study due to DLTs, the other 2 were re-dosed at 3 mg)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/m
Arm/Group | Part A1-1 mg RO7119929 | Part A1-3 mg RO7119929 | Part A1 -4 mg RO7119929 | Part A1 - 6 mg RO7119929 | Part A1 -9 mg RO7119929 | Part B1-5 mg RO7119929
Number analyzed (Participants) | 4 | 6 | 3 | 10 | 4 | 18
ng/m
  Cycle 1, after 1st dose (Prodrug) | 1.29 (146) | 1.94 (46.8) | 1.85 (62.1) | 2.34 (90.6) | 3.67 (178) | 3.18 (204)
  Cycle 1, after 1st dose (Active Drug) | 7.35 (37.4) | 25.1 (49.0) | 39.7 (7.89) | 48.4 (64.0) | 60.9 (16.3) | 49.9 (40.2)
  Cycle 2, after 4th dose (Prodrug): number analyzed (Participants) | 4 | 6 | 3 | 10 | 0 | 18
  Cycle 2, after 4th dose (Prodrug) | 1.46 (231) | 2.49 (21.4) | 2.01 (34.6) | 2.77 (54.9) |  | 4.30 (299)
  Cycle 2, after 4th dose (Active Drug): number analyzed (Participants) | 4 | 6 | 3 | 10 | 0 | 18
  Cycle 2, after 4th dose (Active Drug) | 7.28 (40.5) | 26.3 (52.8) | 30.7 (26.8) | 44.7 (92.7) |  | 50.2 (32.7)

4. Secondary Outcome: Maximum Concentration (Cmax) for RO7119929 Following Administration of RO7119929, Oral Step-Up Dose
Time Frame: Cycle 1 Day 15, Cycle 2 Day 1 (Cycle duration is 21 days)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part A2- 2/5/5 mg RO7119929: Participants received RO7119929 QW with a step-up dosing of 2/5/5 mg.
- Part A2- 2/5/6 mg RO7119929: Participants received RO7119929 QW with a step-up dosing of 2/5/6 mg.
Arm/Group | Part A2- 2/5/5 mg RO7119929 | Part A2- 2/5/6 mg RO7119929
Number analyzed (Participants) | 4 | 3
ng/mL
  Prodrug: Cycle 1 Day 15 | 3.49 (116) | 1.97 (181)
  Prodrug: Cycle 2 Day 1 | 2.37 (48.9) | 3.58 (156)
  Active Drug: Cycle 1 Day 15 | 41.1 (54.9) | 39.6 (16.3)
  Active Drug: Cycle 2 Day 1 | 35.9 (52.3) | 44.4 (32.7)

5. Secondary Outcome: Time of Maximum Concentration Observed (Tmax) for RO7119929 Following Administration of RO7119929
Time Frame: Cycle 1, after 1st dose, Cycle 2, after 4th dose (Each cycle is 21 days)
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Part A1-1 mg RO7119929 | Part A1-3 mg RO7119929 | Part A1 -4 mg RO7119929 | Part A1 - 6 mg RO7119929 | Part A1 -9 mg RO7119929 | Part B1-5 mg RO7119929
Number analyzed (Participants) | 4 | 6 | 3 | 10 | 4 | 18
hour
  Cycle 1, after 1st dose (Prodrug) | 1.02 [0.48 to 4.22] | 1.50 [0.47 to 4.02] | 1.02 [0.53 to 1.08] | 1.53 [0.50 to 3.17] | 1.28 [0.50 to 2.15] | 1.54 [0.52 to 4.07]
  Cycle 1, after 1st dose (Active Drug) | 2.14 [1.03 to 4.22] | 2.07 [1.43 to 5.03] | 1.52 [1.02 to 1.53] | 2.00 [0.97 to 4.03] | 1.83 [1.52 to 2.15] | 3.01 [1.00 to 6.50]
  Cycle 2, after 4th dose (Prodrug): number analyzed (Participants) | 4 | 6 | 3 | 10 | 0 | 18
  Cycle 2, after 4th dose (Prodrug) | 1.03 [0.33 to 3.03] | 0.79 [0.25 to 2.83] | 1.53 [0.53 to 4.03] | 1.08 [0.55 to 3.07] |  | 1.17 [0.53 to 4.02]
  Cycle 2, after 4th dose (Active Drug): number analyzed (Participants) | 4 | 6 | 3 | 10 | 0 | 18
  Cycle 2, after 4th dose (Active Drug) | 2.28 [1.03 to 3.75] | 1.74 [1.17 to 4.12] | 1.53 [1.08 to 4.03] | 1.55 [1.08 to 5.85] |  | 2.17 [1.50 to 4.13]

6. Secondary Outcome: Time of Maximum Concentration Observed (Tmax) for RO7119929 Following Administration of RO7119929, Oral Step-Up Dose
Time Frame: Cycle 1 Day 15, Cycle 2 Day 1 (Cycle duration is 21 days)
Measure: Median (Full Range); unit: hours
Arm/Group | Part A2- 2/5/5 mg RO7119929 | Part A2- 2/5/6 mg RO7119929
Number analyzed (Participants) | 4 | 3
hours
  Prodrug: Cycle 1 Day 15 | 0.51 [0.25 to 0.98] | 1.02 [0.5 to 2.08]
  Prodrug: Cycle 2 Day 1 | 0.78 [0.42 to 2.07] | 2.35 [1.45 to 3.05]
  Active Drug: Cycle 1 Day 15 | 1.03 [0.85 to 1.50] | 1.98 [1.30 to 3.22]
  Active Drug: Cycle 2 Day 1 | 1.43 [1.00 to 2.07] | 2.35 [1.98 to 3.05]

7. Secondary Outcome: Area Under the Curve (AUC) for RO7119929 Following Administration of RO7119929
Time Frame: Cycle 1, after 1st dose, Cycle 2, after 4th dose (Each cycle is 21 days)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part A1-1 mg RO7119929 | Part A1-3 mg RO7119929 | Part A1 -4 mg RO7119929 | Part A1 - 6 mg RO7119929 | Part A1 -9 mg RO7119929 | Part B1-5 mg RO7119929
Number analyzed (Participants) | 4 | 6 | 3 | 10 | 4 | 18
ng*hr/mL
  Cycle 1, after 1st dose (Prodrug): number analyzed (Participants) | 2 | 6 | 3 | 10 | 4 | 18
  Cycle 1, after 1st dose (Prodrug) | 6.27 (46.0) | 4.94 (52.6) | 3.52 (41.0) | 6.55 (71.6) | 8.93 (141) | 1.17 (71.6)
  Cycle 1, after 1st dose (Active Drug) | 31.4 (50.7) | 123 (41.6) | 164 (4.51) | 251 (69.9) | 314 (28.3) | 265 (48.9)
  Cycle 2, after 4th dose (Prodrug): number analyzed (Participants) | 2 | 6 | 3 | 10 | 0 | 18
  Cycle 2, after 4th dose (Prodrug) | 7.91 (43.5) | 6.08 (18.8) | 4.79 (127) | 6.82 (46.3) |  | 10.8 (261)
  Cycle 2, after 4th dose (Active Drug): number analyzed (Participants) | 4 | 6 | 3 | 10 | 0 | 18
  Cycle 2, after 4th dose (Active Drug) | 39.9 (57.4) | 130 (42.9) | 155 (6.28) | 202 (56.0) |  | 242 (32.8)

8. Secondary Outcome: Area Under the Curve (AUC) for RO7119929 Following Administration of RO7119929, Oral Step-Up Dose
Time Frame: Cycle 1 Day 15, Cycle 2 Day 1 (Cycle duration is 21 days)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part A2- 2/5/5 mg RO7119929 | Part A2- 2/5/6 mg RO7119929
Number analyzed (Participants) | 4 | 3
ng*hr/mL
  Prodrug: Cycle 1 Day 15 | 5.38 (89.6) | 4.79 (134)
  Prodrug: Cycle 2 Day 1 | 5.01 (73.9) | 8.04 (167)
  Active Drug: Cycle 1 Day 15 | 213 (31.1) | 170 (23.5)
  Active Drug: Cycle 2 Day 1 | 178 (24.1) | 214 (21.4)

9. Secondary Outcome: Half-Life (T1/2) for RO7119929 Following Administration of RO7119929
Time Frame: Cycle 1, after 1st dose, Cycle 2, after 4th dose (Each cycle is 21 days)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part A1-1 mg RO7119929 | Part A1-3 mg RO7119929 | Part A1 -4 mg RO7119929 | Part A1 - 6 mg RO7119929 | Part A1 -9 mg RO7119929 | Part B1-5 mg RO7119929
Number analyzed (Participants) | 4 | 6 | 3 | 10 | 4 | 18
hours
  Cycle 1, after 1st dose (Prodrug): number analyzed (Participants) | 2 | 6 | 3 | 10 | 4 | 18
  Cycle 1, after 1st dose (Prodrug) | 0.896 (3.77) | 1.54 (31.1) | 1.02 (22.7) | 1.84 (58.3) | 2.46 (65.0) | 1.70 (35.3)
  Cycle 1, after 1st dose (Active Drug) | 3.23 (48.8) | 4.74 (24.9) | 6.3 (26.1) | 5.35 (43.8) | 4.85 (14.2) | 4.86 (35.5)
  Cycle 2, after 4th dose (Prodrug): number analyzed (Participants) | 2 | 6 | 3 | 10 | 0 | 18
  Cycle 2, after 4th dose (Prodrug) | 1.45 (30.3) | 1.33 (37.7) | 1.38 (75.0) | 1.55 (55.5) |  | 1.45 (61.8)
  Cycle 2, after 4th dose (Active Drug): number analyzed (Participants) | 4 | 6 | 3 | 10 | 0 | 18
  Cycle 2, after 4th dose (Active Drug) | 3.74 (37.6) | 4.93 (14.9) | 5.12 (16.9) | 5.00 (16.4) |  | 3.89 (19.0)

10. Secondary Outcome: Half-Life (T1/2) for RO7119929 Following Administration of RO7119929, Oral Step-Up Dose
Time Frame: Cycle 1 Day 15, Cycle 2 Day 1 (Cycle duration is 21 days)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part A2- 2/5/5 mg RO7119929 | Part A2- 2/5/6 mg RO7119929
Number analyzed (Participants) | 4 | 3
hours
  Prodrug: Cycle 1 Day 15 | 1.49 (42.4) | 1.56 (57.4)
  Prodrug: Cycle 2 Day 1 | 1.40 (27.8) | 1.53 (74.5)
  Active Drug: Cycle 1 Day 15 | 5.11 (24.6) | 5.84 (14.5)
  Active Drug: Cycle 2 Day 1 | 5.62 (20.8) | 6.11 (28.9)

11. Secondary Outcome: Progression-Free Survival (PFS) According to RECIST v1.1
Description: Progression-free survival (PFS) is defined as the time from randomization to disease progression or death from any cause.
Time Frame: Baseline up to approximately 14 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A1-1 mg RO7119929 | Part A1-3 mg RO7119929 | Part A1 -4 mg RO7119929 | Part A1 - 6 mg RO7119929 | Part A1 -9 mg RO7119929 | Part B1-5 mg RO7119929 | Part A2- 2/5/5 mg RO7119929 | Part A2- 2/5/6 mg RO7119929 | Part A3-4 mg RO7119929
Number analyzed (Participants) | 4 | 6 | 3 | 10 | 4 | 18 | 4 | 5 | 1
Months | 1.2 [1.2 to NA] — In the chosen method to calculate the 95% confidence interval, the upper bound is not found | 1.4 [1.2 to 1.4] | 2.8 [1.2 to NA] — In the chosen method to calculate the 95% confidence interval, the upper bound is not found | 1.4 [1.3 to 2.8] | 1.2 [1.2 to NA] — In the chosen method to calculate the 95% confidence interval, the upper bound is not found | 1.6 [1.2 to 2.4] | 2.7 [2.4 to NA] — In the chosen method to calculate the 95% confidence interval, the upper bound is not found | 2.8 [1.2 to NA] — In the chosen method to calculate the 95% confidence interval, the upper bound is not found | 3.9 [3.9 to 3.9]

12. Secondary Outcome: Objective Response Rate (ORR) According to RECIST v1.1
Description: ORR is defined as the number of patients who achieve a response, which can either be complete response (complete disappearance of lesions) or partial response (reduction in the sum of maximal tumor diameters by at least 30% or more).
Time Frame: Baseline up to approximately 14 months
Population: Participants with missing tumor assessments and were not included in the efficacy analysis population for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Part A1-1 mg RO7119929 | Part A1-3 mg RO7119929 | Part A1 -4 mg RO7119929 | Part A1 - 6 mg RO7119929 | Part A1 -9 mg RO7119929 | Part B1-5 mg RO7119929 | Part A2- 2/5/5 mg RO7119929 | Part A2- 2/5/6 mg RO7119929 | Part A3-4 mg RO7119929
Number analyzed (Participants) | 4 | 6 | 3 | 9 | 3 | 18 | 4 | 4 | 1
Participants
  Complete Response | 0 [0 to 62.24] | 0 [0 to 45.93] | 0 [0 to 70.76] | 1 [0.28 to 48.25] | 0 [0 to 70.76] | 0 [0 to 18.53] | 0 [0 to 60.24] | 0 [0 to 60.24] | 0 [0 to 97.50]
  Partial Response | 0 [0 to 62.24] | 0 [0 to 45.93] | 0 [0 to 70.76] | 0 [0 to 33.63] | 0 [0 to 70.76] | 0 [0 to 18.53] | 0 [0 to 60.24] | 0 [0 to 60.24] | 0 [0 to 97.50]

13. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from randomization to death
Time Frame: Baseline up to approximately 14 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A1-1 mg RO7119929 | Part A1-3 mg RO7119929 | Part A1 -4 mg RO7119929 | Part A1 - 6 mg RO7119929 | Part A1 -9 mg RO7119929 | Part B1-5 mg RO7119929 | Part A2- 2/5/5 mg RO7119929 | Part A2- 2/5/6 mg RO7119929 | Part A3-4 mg RO7119929
Number analyzed (Participants) | 4 | 6 | 3 | 10 | 4 | 18 | 4 | 5 | 1
Months | 3.2 [1.6 to NA] — In the chosen method to calculate the 95% confidence interval, the upper bound is not found | 5.1 [2.9 to NA] — In the chosen method to calculate the 95% confidence interval, the upper bound is not found | 7.9 [5.5 to NA] — In the chosen method to calculate the 95% confidence interval, the upper bound is not found | NA [5.5 to NA] — In the chosen method to calculate the 95% confidence interval, the upper bound is not found | 2.9 [2.9 to NA] — In the chosen method to calculate the 95% confidence interval, the upper bound is not found | 8.0 [3.9 to NA] — In the chosen method to calculate the 95% confidence interval, the upper bound is not found | NA [3.4 to NA] — In the chosen method to calculate the 95% confidence interval, the upper bound is not found | NA [NA to NA] — In the chosen method to calculate the 95% confidence interval, the upper bound is not found | NA [NA to NA] — In the chosen method to calculate the 95% confidence interval, the upper bound is not found

ADVERSE EVENTS:
Time Frame: Baseline up to 14 months
Description: Number of events includes all occurrences
Groups:
- Part A1-6 mg RO7119929: Participants received 6 mg RO7119929 every week in 3-week cycles
- Part A1-9 mg RO7119929: Participants received 9 mg RO7119929 every week in 3-week cycles
Arm/Group | Part A1-1 mg RO7119929 | Part A1-3 mg RO7119929 | Part A1 -4 mg RO7119929 | Part A1-6 mg RO7119929 | Part A1-9 mg RO7119929 | Part B1-5 mg RO7119929 | Part A2- 2/5/5 mg RO7119929 | Part A2- 2/5/6 mg RO7119929 | Part A3-4 mg RO7119929
All-Cause Mortality (participants affected / at risk) | 3/4 | 4/6 | 2/3 | 4/10 | 4/4 | 8/18 | 1/4 | 0/5 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/6 | 2/3 | 4/10 | 4/4 | 11/18 | 1/4 | 2/5 | 0/1
Other Adverse Events (participants affected / at risk) | 3/4 | 6/6 | 3/3 | 10/10 | 3/4 | 18/18 | 4/4 | 5/5 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A1-1 mg RO7119929 (N=4) | Part A1-3 mg RO7119929 (N=6) | Part A1 -4 mg RO7119929 (N=3) | Part A1-6 mg RO7119929 (N=10) | Part A1-9 mg RO7119929 (N=4) | Part B1-5 mg RO7119929 (N=18) | Part A2- 2/5/5 mg RO7119929 (N=4) | Part A2- 2/5/6 mg RO7119929 (N=5) | Part A3-4 mg RO7119929 (N=1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 2 (2) | 2 (6) | 4 (4) | 4 (4) | 9 (11) | 0 (0) | 2 (3) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A1-1 mg RO7119929 (N=4) | Part A1-3 mg RO7119929 (N=6) | Part A1 -4 mg RO7119929 (N=3) | Part A1-6 mg RO7119929 (N=10) | Part A1-9 mg RO7119929 (N=4) | Part B1-5 mg RO7119929 (N=18) | Part A2- 2/5/5 mg RO7119929 (N=4) | Part A2- 2/5/6 mg RO7119929 (N=5) | Part A3-4 mg RO7119929 (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (5) | 0 (0) | 3 (8) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (4) | 0 (0) | 1 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (19) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (8) | 0 (0) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 6 (17) | 3 (5) | 7 (80) | 1 (1) | 14 (43) | 3 (10) | 3 (12) | 1 (2)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (6) | 1 (1) | 5 (6) | 0 (0) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Procalcitonin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/85/NCT04338685/Prot_SAP_000.pdf